CLINICAL TRIAL: NCT05707403
Title: Investigation of Pharmacokinetics and Absolute Oral Bioavailability of BI 1015550 Administered as an Oral Dose With an Intravenous Microtracer Dose of [14C]-BI 1015550 in Healthy Male Volunteers
Brief Title: A Study in Healthy Men to Test How BI 1015550 is Taken up and Handled by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0030; 2022-003119-27 (EudraCT Number)
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test treatment (T) followed by Reference treatment (R) (Experimental)
  Interventions: Drug: BI 1015550; Drug: BI 1015550 mixed with [C-14]-BI 1015550

INTERVENTIONS:
Drug: BI 1015550 — Treatment T
  Other Names: Nerandomilast; JASCAYD®
Drug: BI 1015550 mixed with [C-14]-BI 1015550 — Treatment R
  Other Names: Nerandomilast; JASCAYD®

SUMMARY:
This trial is intended to examine the absolute oral bioavailability of BI 1015550 as tablet formulation for oral administration, using an intravenous microtracer approach with [14C]-labelled BI 1015550. These data are considered necessary to further support the understanding of the pharmacokinetics of BI 1015550.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 40 to 100 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders (including but not limited to major depressive disorder or history of suicide attempts)
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ICON, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A non-randomised, open-label, single period, single arm trial to determine the absolute oral bioavailability of BI 1015550 in healthy male subjects.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 18 mg BI 1015550 / 100 μg BI 1015550 (C-14): One film-coated tablet of 18 milligram (mg) BI 1015550 was administered as single oral dose with 240 milliliter of water after an overnight fast of at least 10 hours on Day 1 as test treatment (T). 100 microgram (μg) BI 1015550 (C-14) solution (consisting of 90 μg unlabelled BI 1015550 mixed with 10 μg labelled [14C]-BI 1015550 in 10 mL intravenous solution with a final concentration of 10 μg BI 1015550 (C-14)/mL) was administered as single intravenous infusion over 15 minutes on Day 1 as reference treatment (R). The radioactive dose per infusion was ~40 kilobecquerel (kBq).
Period: Overall Study
Arm/Group | 18 mg BI 1015550 / 100 μg BI 1015550 (C-14)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All subjects who were treated with at least one dose of trial drug.
Arm/Group | 18 mg BI 1015550 / 100 μg BI 1015550 (C-14)
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.9 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Dose Normalized Area Under the Concentration-time Curve of BI 1015550 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: Dose normalized AUC0-inf of [14C]-BI 1015550 after intravenous (i.v.) administration and AUC0-inf of BI 1015550 after oral (p.o.) administration are reported. The analysis was performed only on the pharmacologically active R-enantiomer.
Time Frame: Between waking up and still prior to drug intake and 0.5*, 0.75*, 1*, 1.5*, 1.58±, 1.67±, 1.75, 2, 2.5±, 3, 4, 5±, 6, 7±, 8, 12, 16, 24, 36, 48, 72, 120, 168, 216± hours after intake of oral BI 1015550 tablet, *for T treatment, ±only for R treatment.
Population: Pharmacokinetic (PK) set (PKS): All subjects in the treated set (TS) who provided at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to non-evaluability.
Measure: Geometric Mean (Standard Error); unit: Hours*millimole/liter/kilogram
Groups:
- R-BI 1015550 18 mg tablet (T): Unlabelled pharmacologically active R-enantiomer of one film-coated tablet of 18 mg BI 1015550, as test treatment (T).
- 14C-R-BI 1015550 10 μg i.v. (R): Intravenous microtracer infusion of 100 ug BI 1015550 (C-14) solution containing 10 ug 14C radiolabelled pharmacologically active R-enantiomer of BI 1015550, as reference treatment (R).
Arm/Group | R-BI 1015550 18 mg tablet (T) | 14C-R-BI 1015550 10 μg i.v. (R)
Number analyzed (Participants) | 8 | 8
Hours*millimole/liter/kilogram | 118.27 (1.07) | 161.69 (1.07)
Statistical Analysis 1: Comparison: R-BI 1015550 18 mg tablet (T) vs 14C-R-BI 1015550 10 μg i.v. (R); Analysis of variance (ANOVA) model on the logarithmic scale. That is, the PK endpoints were logtransformed (natural logarithm) prior to fitting the ANOVA model and then then back-transformed to the original scale to provide the point estimate and 90% confidence interval. The model included effects accounting for the following sources of variation: 'subjects' and 'formulation'. The effect 'subjects' was considered as random, whereas the 'formulation' effect was considered as fixed; Test type: Other; Ratio (T/R) [%] = 73.15, 90% CI 2-sided [67.32 to 79.48] — Ratio [%] is calculated as Test / Reference Intra-individual geometric Coefficient of Variation (gCV) = 8.8 %

2. Secondary Outcome: Dose Normalized Maximum Measured Concentration of BI 1015550 in Plasma (Cmax)
Description: Dose normalized Cmax of BI 1015550 after oral administration and Cmax of [14C]-BI 1015550 after intravenous administration is reported. The analysis was performed only on the pharmacologically active R-enantiomer.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomole/Liter/microgram
Arm/Group | R-BI 1015550 18 mg tablet (T) | 14C-R-BI 1015550 10 μg i.v. (R)
Number analyzed (Participants) | 8 | 8
Picomole/Liter/microgram | 24.53 (1.13) | 73.05 (1.13)
Statistical Analysis 1: Comparison: R-BI 1015550 18 mg tablet (T) vs 14C-R-BI 1015550 10 μg i.v. (R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio (T/R) [%] = 33.58, 90% CI 2-sided [29.40 to 38.36] — Ratio [%] is calculated as Test / Reference Intra-individual geometric Coefficient of Variation (gCV) = 14.1 %

ADVERSE EVENTS:
Time Frame: For all-cause mortality: From study start until end of study up to 22 days. For serious and other adverse events: From drug administration until the last dose, plus 7 days of residual effect period, up to 7 days.
Description: Treated Set (TS): All subjects who were treated with at least one dose of trial drug.
Arm/Group | 18 mg BI 1015550 / 100 μg BI 1015550 (C-14)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT05707403/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT05707403/SAP_001.pdf